CLINICAL TRIAL: NCT01764087
Title: An Open-label Phase I/II Study of KX2-391 in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: A Study of KX2-391 With Paclitaxel in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-KXI-101
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2014-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Gastric Cancer; Breast Cancer
Keywords: Stomach Neoplasms; Breast Neoplasms; Carcinoma; Neoplasms; Paclitaxel; Tubulin Modulators; Antimitotic Agents; Protein Kinase Inhibitors; Enzyme Inhibitors; Pharmacologic Actions
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Carcinoma; Neoplasms | interventions — tirbanibulin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KX2-391 and Paclitaxel (Experimental): The phase I portion is a standard, three-patient per cohort, dose escalation schedule will be used. 3 or 6 subjects with solid tumor per dose group will likely be necessary to determine the MTD of KX2-391 in combination with weekly paclitaxel. With paclitaxel dose fixed at 80 mg/m2/weekly, KX2-391 treatment will be started at 20 mg dose once daily (QD)
  The phase II portion of this trial has a design to determine the efficacy of KX2-391 when administered in combination with paclitaxel in 20 subjects with stomach cancer and 20 subjects with breast cancer
  Interventions: Drug: KX2-391 and Paclitaxel

INTERVENTIONS:
Drug: KX2-391 and Paclitaxel — A treatment cycle in phase I will consist of 28 days, according to the following schedule:
  KX2-391 20 mg PO once daily, Weekly paclitaxel 80 mg/m2 given intravenously over 1 hour on day 1, 8, and 15 of a 28 day cycle.
  The trial will initially test the combination of weekly paclitaxel and KX2-391 given PO, once daily , continuously. In case of 2 dose-limiting toxicities (DLT) in the first cohort, this intervention will be terminated
  A treatment cycle in phase II will consist of 28 days, according to the following schedule:
  KX2-391 MTD PO once daily, Weekly paclitaxel 80 mg/m2 given intravenously over 1 hour on day 1, 8, and 15 of a 28 day cycle.
  Other Names: KX01; Taxol

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) of KX2-391 in Combination with paclitaxel in Phase I, and to evaluate the efficacy of KX2-391 in combination with paclitaxel in patients who are diagnosed as gastric and breast cancer, respectively in Phase II.

ELIGIBILITY:
Inclusion Criteria:

Phase I Portion:

- Diagnosis of solid tumors on histopathological examination or cytological examination for which no standard of care is available or conventional treatment modalities have no therapeutic effect at the time of entering into the study

Phase II Portion:

* Diagnosis of advanced/metastatic/recurrent stomach cancer or breast cancer on histopathological examination or cytological examination for which no standard of care is available or conventional treatment modalities have no therapeutic effect at the time of entering into the study
* Subjects with stomach cancer without prior taxane therapy
* Subjects with breast cancer with prior taxane therapy
* (Optional) Providing exploratory biomarker informed consent form to obtain archival tumor tissue and/or new tumor biopsy sample

Common:

1. Based on clinical screening,

   ① If radiotherapy was given, at least 4 weeks should have passed from the last treatment date and the patient should have recovered from the toxicity (However, for limited regional radiotherapy, at least 2 weeks from the last treatment date)

   ② If hormonal therapy was given, at least 2 weeks should have passed from the last treatment date and the patient should have recovered from the toxicity.

   ③ If chemotherapy was given, at least 3 weeks should have passed from the last treatment date and the patient should have recovered from the toxicity (However, for nitrosourea or mitomycin, at least 6 weeks)
2. Aged ≥ 20 years
3. ECOG (Eastern Cooperative Oncology Group) ≤ 2
4. Life expectancy ≥ 12 weeks
5. Should meet the followings,

   ① Bone marrow function ANC (Absolute Neutrophil Count) ≥ 1.5 X 109/L, PLT (Platelet Count) ≥ 100 X 109/L, Hemoglobin ≥ 9.0 g/dl (In the case of hemoglobin of < 9.0 g/dl, the patient can be enrolled if the value is reversed to ≥ 9.0 g/dl.)

   ② Kidney function Creatinine Clearance > 50 ml/min or Serum Clearance ≤ 1.5 mg/dl

   ③ Liver function AST (Aspartate Aminotransferase)/ALT (Alanine Aminotransferase)/ALP (Alkaline Phosphatase) ≤ 3.0 X UNL and Total bilirubin ≤ 2.0 mg/dl (With bone metastasis, ALP ≤ 5.0 X UNL)
6. At least one measurable lesions with the length of the longest diameter of ≥ 10 mm on spiral CT or multidetector CT or ≥ 20 mm on conventional CT
7. Subjects who voluntarily consent to participate in this study and sign the written informed consent form

Exclusion Criteria:

1. Uncontrolled central nervous system metastasis
2. Malignant ascites requiring surgical treatment
3. Subjects who have blood malignancies including leukemia; or who have received or will receive bone marrow transplantation
4. Severe concurrent diseases as follows,

   ① History of unstable angina, heart failure, atrial or ventricular arrhythmia requiring pharmacological treatment, or having received treatment for myocardial infarction within 6 months (however, may be included under the judgment of the investigator if medically controlled), heart failure of Class III or IV by New York Heart Association Classes, or left ventricular ejection fraction of < 40%

   ② Receiving therapeutic dose administration of coumarin-type anticoagulants (however, up to 2 mg daily is permitted for line opening)

   ③ Uncontrolled diabetes (fasting plasma glucose > 2.0 X UNL), severe hypertension, thyroid disorder and active infectious disease

   ④ Psychiatric or neurological history including dementia or epilepsy which may threaten the compliance with this protocol

   ⑤ A condition not allowing oral application of tablet formulation, and any clinically significant gastrointestinal abnormalities which may interfere with taking, passing or absorption of the study drug
5. Using disallowed concomitant medications (strong CYP3A4 (Cytochrome P450 3A4) inhibitors or inducers) (When a patient is using any of the disallowed concomitant medications below, wash-out of 1 week from the medication date is required)
6. Received other investigational product within 4 weeks prior to the administration of this study drug
7. Pregnant or breast-feeding women (however, women with 12 months of natural (spontaneous) amenorrhea or surgical bilateral oophorectomy (alone or with hysterectomy) at least 6 weeks ago, with appropriate clinical profile (e.g., appropriate age, history of vasomotor symptoms), will be considered women postmenopausal and of non-childbearing potential. In the case of oophorectomy alone, a woman will be considered to be of non-childbearing potential only if her reproductive condition is confirmed by follow-up hormone level assessment)
8. History of hypersensitivity to paclitaxel, compounds with similar chemical structure, or cremophor (polyoxyethylated castor oil) ingredient
9. Neuropathy of grade ≥ 3 based on clinical screening
10. Known history of hepatitis B or C and known history of HIV serum positive
11. Others unable to participate in the study under the judgment of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) in Phase I Portion | From start of the treatment to end of cycle 1, which are 4 weeks
  Maximum tolerated dose (MTD) of KX2-391 in combination with weekly paclitaxel as determined by number of participants With DLTs related to KX2-391 in combination with weekly paclitaxel
Tumor Overall Response Rates (ORRs) in Phase II Portion | In every 2 cycles up to end of the treatment, an expected average of 16 weeks
  The efficacy (overall response rate; ORR; complete response (CR) + partial response (PR)) of KX2-391 in combination with weekly paclitaxel at the MTD established during the phase I portion of this trial based on Response Evaluation Criteria in Solid Tumor (RECIST) 1.1

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Evaluation in Phase I Portion | Time points at day 0, 1 and 8 in cycle 1
  PK parameters, including but not limited to, plasma concentration, AUC (Area Under Curve) 0-t, Cmax, Tmax, and T1/2 of KX2-391 alone and in combination with weekly paclitaxel
The Preliminary Efficacy Data in Phase I Portion | In every 2 cycles up to end of the treatment, an expected average of 8 weeks
  The preliminary efficacy of KX2-391 in combination with weekly paclitaxel as determined by ORRs based on RECIST 1.1
Safety in Phase II Portion | From start of the treatment to end of the treatment, an expected average of 16 weeks
  Adverse events and their frequency, duration and severity, physical examination, laboratory parameters, vital signs and ECG change monitoring as determined based on CTCAE (Common Toxicity Criteria for Adverse Effects) 4.03
The Efficacy Data in Phase II Portion | Up to die, an expected average of 24 weeks
  Overall survival (OS), progression free survival (PFS), time to tumor progression (TTP) and duration of response
Pharmacokinetic (PK) Evaluation in Phase II Portion | Time points at day 1 and 8 in cycle 1
  PK parameters, including but not limited to, plasma concentration, AUC0-t, Cmax, Tmax, and T1/2 of KX2-391 alone and in combination with weekly paclitaxel

OTHER OUTCOMES:
Pharmacodynamic (PD) Evaluation in Phase I Portion | Time points at day 0 and 1 in cycle 1
  Pre-dose and post-dose tubulin inhibition in peripheral blood monocytes extracted from blood samples, as measured by immunofluorescence staining
Exploratory Biomarker Evaluation in Phase II Portion | Time points at day -6 and day 0
  Pre-dose and post-dose Src signaling inhibition (p-Src and Ki-67) in archival tumor tissue and new biopsy sample, as measured by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul